CLINICAL TRIAL: NCT04354428
Title: Efficacy of Novel Agents for Treatment of SARS-CoV-2 Infection Among High-Risk Outpatient Adults: An Adaptive Randomized Platform Trial
Brief Title: Treatment for COVID-19 in High-Risk Adult Outpatients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low number of events contributing to primary outcome
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Christine Johnston, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009878; INV-017062 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Outpatient; Treatment; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid; Hydroxychloroquine; Azithromycin; Folic Acid; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Ascorbic acid and Folic acid (Placebo Comparator): Ascorbic acid 500 mg orally twice on Day 1, followed by 250 mg orally twice daily for 9 days + folic acid 800 µg orally once on Day 1, followed by 400 µg orally once daily for an additional 4 days (Days 2 to 5)
  Interventions: Drug: Ascorbic Acid; Drug: Folic Acid
- Hydroxychloroquine and Folic Acid (Experimental): HCQ 400 mg orally twice on Day 1, followed by 200 mg orally twice daily for an additional 9 days (Days 2 to 10) + placebo (folic acid 800 µg orally once on Day 1, followed by 400 µg orally once daily for an additional 4 days [Days 2 to 5])
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Folic Acid
- Hydroxychloroquine and Azithromycin (Experimental): HCQ 400 mg orally twice on Day 1, followed by 200 mg orally twice daily for an additional 9 days (Days 2 to 10) + azithromycin 500 mg orally once on Day 1, followed by 250 mg orally once daily for an additional 4 days (Days 2 to 5).
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Azithromycin
- Lopinavir-ritonavir (Experimental): LPV/r 800 mg-200 mg orally twice on Day 1, followed by 400 mg 100 mg orally twice daily for an additional 9 days (Days 2 to 10)
  Interventions: Drug: Lopinavir 200 MG / Ritonavir 50 MG [Kaletra]
- Ascorbic acid (Placebo Comparator): Ascorbic acid 1 gm orally twice on Day 1, followed by 500 mg orally twice daily for 9 days
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Eligible participants in a household randomized to this study arm will receive ascorbic acid only or ascorbic acid and additional drug therapy
  Other Names: Placebo
  Arms: Ascorbic acid; Ascorbic acid and Folic acid
Drug: Hydroxychloroquine Sulfate — Eligible participants in a household randomized to this study arm will receive hydrochloroquine and folic acid therapy
  Other Names: Intervention A
  Arms: Hydroxychloroquine and Azithromycin; Hydroxychloroquine and Folic Acid
Drug: Azithromycin — Eligible participants in a household randomized to this study arm will receive hydrochloroquine and azithromycin therapy
  Other Names: Intervention B
  Arms: Hydroxychloroquine and Azithromycin
Drug: Folic Acid — Eligible participants in a household will receive folic acid and an additional intervention drug
  Other Names: Placebo
  Arms: Ascorbic acid and Folic acid; Hydroxychloroquine and Folic Acid
Drug: Lopinavir 200 MG / Ritonavir 50 MG [Kaletra] — Eligible participants in a household randomized to this study arm will receive lopinavir-ritonavir therapy
  Other Names: Intervention C
  Arms: Lopinavir-ritonavir

SUMMARY:
This is a randomized trial for the treatment of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection in high-risk adults not requiring hospital admission.The overarching goal of this study is to assess the effectiveness of interventions on the incidence of lower respiratory tract infection (LRTI) progression among high-risk adult outpatients with SARS-CoV-2 infection to inform public health control strategies.

DETAILED DESCRIPTION:
This is a randomized, multi-center, placebo-equivalent (ascorbic acid + folic acid)-controlled, blinded platform trial. Eligible participants will be enrolled and randomized to Hydrocychloroquine (HCQ) + placebo (folic acid), HCQ + azithromycin, lopinavir-ritonavir (LPV/r) or placebo (ascorbic acid + folic acid). Initially, this study will enroll up to 495 eligible adults ( with high risk for Lower respiratory tract infection (LRTI) progression at baseline who are PCR-confirmed SARS-CoV-2 infection (165 per arm). An additional cohort of 135 eligible adults without risk factors for LRTI progression at baseline who are PCR-confirmed SARS-CoV-2 infection will be enrolled for the co-primary virologic outcome. During the 28 study days, participants will take the medication, complete surveys, collect mid nasal swab for viral quantification, and assess symptoms for progression to LRTI. Additional arms will be added should new potential agents be discovered or combination treatments be proposed. In addition, arms may be dropped prior to completion if deemed futile or if there is a safety signal.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 80 years of age, inclusive, at the time of signing the informed consent
* Willing and able to provide informed consent
* Laboratory confirmed SARS-CoV-2 infection, with test results within past 72 hours
* COVID-19 symptoms, based on the following criteria: At least TWO of the following symptoms: Fever (≥ 38ºC), chills, rigors, myalgia, headache, sore throat, new olfactory and taste disorder(s), OR o At least ONE of the following symptoms: cough, shortness of breath or difficulty breathing (Lopinavir-Ritonavir Platform)
* Access to device and internet for Telehealth visits
* At increased risk of developing severe COVID-19 disease (at least one of the following)

  1. Age ≥60 years
  2. Presence of pulmonary disease, specifically moderate or severe persistent asthma, chronic obstructive pulmonary disease, pulmonary hypertension, emphysema
  3. Diabetes mellitus (type 1 or type 2), requiring oral medication or insulin for treatment
  4. Hypertension, requiring at least 1 oral medication for treatment
  5. Immunocompromised status due to disease (e.g., those living with human immunodeficiency virus with a CD4 T-cell count of <200/mm3)
  6. Immunocompromised status due to medication (e.g., persons taking 20 mg or more of prednisone equivalents a day, anti-inflammatory monoclonal antibody therapies, or cancer therapies)
  7. Body mass index ≥30 (self-reported)

Exclusion Criteria:

* Known hypersensitivity to HCQ or other 4-aminoquinoline compounds
* Known hypersensitivity to azithromycin or other azalide or macrolide antibiotics
* Currently hospitalized
* Signs of respiratory distress prior to randomization, including respiratory rate >24
* Current medications include HCQ
* Concomitant use of other anti-malarial treatment or chemoprophylaxis
* History of retinopathy of any etiology
* Psoriasis
* Porphyria
* Chronic kidney disease (Stage IV or receiving dialysis)
* Known bone marrow disorders with significant neutropenia (polymorphonuclear leukocytes <1500) or thrombocytopenia (<100 K)
* Concomitant use of digoxin, cyclosporin, cimetidine, amiodarone, or tamoxifen
* Known cirrhosis
* Known personal or family history of long QT syndrome
* History of coronary artery disease with a history of graft or stent
* History of heart failure, Class 2 or greater using the New York Heart Association functional class
* Taking medications associated with prolonged QT and known risk of torsades de points. These medications may include some antipsychotic and antidepressant medications. (Lopinavir-Ritonavir Platform)
* Taking medications associated with prolonged QT such as antipsychotic medications or antidepressants (e.g., citalopram, venlafaxine, and bupropion) and unable to stop during the trial
* Taking warfarin (Coumadin or Jantoven)
* Known history of glucose-6-phosphate-dehydrogenase deficiency
* History of myasthenia gravis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, MPH, Principal Investigator — University of Washington
Locations (6):
- United States (6):
  - Ruth M. Rothstein CORE Center - Cook County Health, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Boston University, Boston, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Washington Coordinating Center, Seattle, Washington
  - UW Virology Research Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study will be made available in accordance with the funder's open access policy.
Supporting Information: Study Protocol, ICF
Time Frame: Within 3 months of publication of primary results.
Access Criteria: De-identified data from the study will be made available in accordance with the funder's open access policy.
URL: https://www.gatesfoundation.org/how-we-work/general-information/open-access-policy

REFERENCES:
- [Derived] Mayfield JJ, Chatterjee NA, Noseworthy PA, Poole JE, Ackerman MJ, Stewart J, Kissinger PJ, Dwyer J, Hosek S, Oyedele T, Paasche-Orlow MK, Paolino K, Friedman PA, Waters C, Moreno J, Leingang H, Heller KB, Morrison SA, Krows ML, Barnabas RV, Baeten J, Johnston C; COVID-19 Early Treatment Team; Sridhar AR. Implementation of a fully remote randomized clinical trial with cardiac monitoring. Commun Med (Lond). 2021 Dec 20;1:62. doi: 10.1038/s43856-021-00052-w. eCollection 2021. PMID 35604806
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Johnston C, Brown ER, Stewart J, Karita HCS, Kissinger PJ, Dwyer J, Hosek S, Oyedele T, Paasche-Orlow MK, Paolino K, Heller KB, Leingang H, Haugen HS, Dong TQ, Bershteyn A, Sridhar AR, Poole J, Noseworthy PA, Ackerman MJ, Morrison S, Greninger AL, Huang ML, Jerome KR, Wener MH, Wald A, Schiffer JT, Celum C, Chu HY, Barnabas RV, Baeten JM; COVID-19 Early Treatment Study Team. Hydroxychloroquine with or without azithromycin for treatment of early SARS-CoV-2 infection among high-risk outpatient adults: A randomized clinical trial. EClinicalMedicine. 2021 Mar;33:100773. doi: 10.1016/j.eclinm.2021.100773. Epub 2021 Feb 27. PMID 33681731

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a remotely conducted study. Participants who completed the informed consent process but did not complete the enrollment process after receiving the study materials are "started" but are not considered to have "completed enrollment". This explains the discrepancy between "Started" and "Completed Enrollment"
Period: Overall Study
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Started | 83 | 71 | 77 | 29 | 29
Completed Enrollment | 80 | 65 | 74 | 27 | 28
Completed | 75 | 62 | 71 | 19 | 25
Not Completed | 8 | 9 | 6 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid | Total
Number analyzed (Participants) | 83 | 71 | 77 | 29 | 29 | 289
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 21 | 19 | 24 | 7 | 8 | 79
  30-39 years | 26 | 28 | 21 | 9 | 9 | 93
  40-49 years | 16 | 13 | 14 | 7 | 6 | 56
  50-59 years | 12 | 5 | 9 | 6 | 3 | 35
  60-69 years | 7 | 5 | 8 | 0 | 2 | 22
  70-80 years | 1 | 1 | 1 | 0 | 1 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex, defined at birth
  Participants
    Female | 45 | 39 | 47 | 17 | 20 | 168
    Male | 38 | 32 | 30 | 12 | 9 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 23 | 18 | 7 | 4 | 82
  Not Hispanic or Latino | 52 | 48 | 59 | 22 | 25 | 206
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 11 | 16 | 0 | 0 | 39
  Asian | 4 | 3 | 4 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 0 | 0 | 3
  Black or African American | 7 | 10 | 9 | 5 | 4 | 35
  White | 41 | 37 | 39 | 18 | 24 | 159
  More than one race | 15 | 10 | 7 | 6 | 0 | 38
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 1 | 4
High Risk [Count of Participants; unit: Participants] — The high risk cohort included participants at increased risk of severe COVID-19 disease based on the following factors (at least one of the following) (see protocol for additional information and definitions):
  1. Age>=60 years
  2. Pulmonary disease, specifically moderate or severe persistent asthma, chronic obstructive pulmonary disease, pulmonary hypertension, emphysema
  3. Diabetes mellitus (Type 1 or Type 2)
  4. Hypertension
  5. Immunocompromised status due to disease
  6. Immunocompromised status due to medication
  7. Body mass index>=30kg/m2 (self-reported)
  Participants | 48 | 37 | 44 | 8 | 10 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Persons With Lower Respiratory Tract Infection (LRTI), Defined as Resting Blood Oxygen Saturation (SpO2<93%) Level Sustained for 2 Readings 2 Hours Apart and Presence of Subjective Dyspnea or Cough
Description: Resting blood oxygen saturation (SpO2<93%) level sustained for 2 readings 2 hours apart and presence of subjective dyspnea or cough
Time Frame: 28 days from enrolment
Population: This outcome was analyzed in the first arm of the platform trial (Ascorbic Acid/Folic Acid HCQ, HCQ/AZ) among the high risk cohort only. The mITT cohort included only those without LRTI at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 47 | 36 | 44 | 29 | 29
Participants | 2 | 0 | 4 | 2 | 1

2. Primary Outcome: Number of Participants With Hospitalization or Mortality
Description: Number of participants with hospitalization or mortality
Time Frame: Day 28 after enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 83 | 71 | 77 | 29 | 29
Participants | 4 | 2 | 3 | 0 | 1

3. Primary Outcome: Time to Clearance of Nasal SARS-CoV-2
Description: Time to clearance of nasal SARS-CoV-2, defined as 2 consecutive negative swabs
Time Frame: Day 1 through Day 14 after enrolment
Population: Included the mITT viral shedding cohort, which includes the mITT cohort participants who do not meet the definition for clearance of viral shedding at baseline (day 1 and 2 swabs negative).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 52 | 49 | 51 | 16 | 21
Days | 7 [6 to 10] | 5 [4 to 6] | 6 [4 to 8] | 4 [3 to NA] — Due to limited participants with events within the followup period, unable to calculate upper confidence interval limit | 5 [3 to 9]

4. Primary Outcome: Time to Resolution of COVID-19 Symptom Resolution in Days
Description: COVID-19 symptoms are based on the following criteria:
  * At least TWO of the following symptoms: Fever (≥ 38ºC), chills, rigors, myalgia, headache, sore throat, new olfactory and taste disorder(s), OR
  * At least ONE of the following symptoms: cough, shortness of breath or difficulty breathing, OR
  * Severe respiratory illness with at least 1 of the following:
    * Clinical or radiological evidence of pneumonia, OR
    * Acute respiratory distress syndrome (ARDS), OR
    * LRTI, defined by resting SpO2<93% sustained for 2 readings 2 hours apart AND presence of subjective dyspnea or cough Death or COVID-19-related hospitalizations will count as a failure to resolve symptoms.
Time Frame: Day 1 through Day 14 after enrolment
Population: mITT Disease Resolution cohort includes participants who meet the COVID-19 disease criteria on day 1. The symptom resolution rate was the primary outcome of the lopinavir-ritonavir adaptive platform arms (lopinavir-ritonavir and ascorbic acid).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 72 | 60 | 65 | 27 | 25
Days | 11.5 [8.5 to NA] — Due to limited participants with events within the followup period, unable to calculate upper confidence interval limit | 10.5 [6.5 to NA] — Due to limited participants with events within the followup period, unable to calculate upper confidence interval limit | NA [9.5 to NA] — Due to limited participants with events within the followup period, unable to calculate median or upper confidence interval limit | NA [NA to NA] — Due to limited participants with events within the followup period, unable to calculate median or confidence interval limit | NA [10.5 to NA] — Due to limited data, unable to calculate Due to limited participants with events within the followup period, unable to calculate median and upper confidence interval limit

5. Secondary Outcome: Number of Participants With Serious Adverse Events and Adverse Events Resulting in Treatment Discontinuation
Description: Serious adverse events (including death and hospitalization) and adverse events resulting in treatment discontinuation
Time Frame: 28 days from enrolment
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 83 | 71 | 77 | 29 | 29
Participants | 6 | 6 | 8 | 9 | 1

6. Secondary Outcome: COVID-19-related Hospitalization Days
Description: Duration of hospitalization among persons who become hospitalized with COVID-19 disease
Time Frame: 28 days from enrolment
Measure: Number; unit: Days
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
Number analyzed (Participants) | 83 | 71 | 77 | 29 | 29
Days | NA — Duration of hospitalization not assessed due to insufficient number of participants with events | NA — Duration of hospitalization not assessed due to insufficient number of participants with events | NA — Duration of hospitalization not assessed due to insufficient number of participants with events | NA — Duration of hospitalization not assessed due to insufficient number of participants with events | NA — Duration of hospitalization not assessed due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: 28 days
Description: Participant reported AE
Arm/Group | Ascorbic Acid and Folic Acid | Hydroxychloroquine and Folic Acid | Hydroxychloroquine and Azithromycin | Lopinavir-ritonavir | Ascorbic Acid
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/71 | 0/77 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/83 | 2/71 | 3/77 | 0/29 | 1/29
Other Adverse Events (participants affected / at risk) | 2/83 | 4/71 | 5/77 | 9/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid and Folic Acid (N=83) | Hydroxychloroquine and Folic Acid (N=71) | Hydroxychloroquine and Azithromycin (N=77) | Lopinavir-ritonavir (N=29) | Ascorbic Acid (N=29)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hemorrhagic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid and Folic Acid (N=83) | Hydroxychloroquine and Folic Acid (N=71) | Hydroxychloroquine and Azithromycin (N=77) | Lopinavir-ritonavir (N=29) | Ascorbic Acid (N=29)
Event leading to treatment discontinuation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4) | 9 (13) | 0 (0)
QT Prolongation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Reaction or Hives

LIMITATIONS AND CAVEATS:
Early termination of HCQ and HCQ/AZ arms as well as lopinavir-ritonavir arms leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol: Hydroxychloroquine and Azithromycin arms (2020-04-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04354428/Prot_002.pdf
  • Study Protocol: Lopinavir-Ritonavir arm (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04354428/Prot_003.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT04354428/SAP_007.pdf
  • Informed Consent Form: Hydroxychloroquine and Azithromycin arms (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT04354428/ICF_004.pdf
  • Informed Consent Form: Lopinavir-Ritonavir arm (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04354428/ICF_005.pdf